CLINICAL TRIAL: NCT01490619
Title: Resilience Promotion in Teens With Type 1 Diabetes: Preventing Negative Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Jill Weissberg-Benchell, Ph.D., Attending Psychologist, Department of Psychiatry, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DK090030-01A1 (NIH)
Record Dates: First submitted 2011-12-07; First posted 2011-12-13 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Adolescent; Resilience; Prevention; Depression
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Thinking in Teens (Experimental): Group-based, manualized program, based on cognitive behavioral therapy techniques.
  Interventions: Behavioral: Healthy Thinking In Teens
- Advanced Diabetes Education (Active Comparator): Group-based, manualized program designed to provide diabetes education, focused on adolescent-specific topics.
  Interventions: Other: Advanced Diabetes Education.

INTERVENTIONS:
Behavioral: Healthy Thinking In Teens — 9 sessions. Manualized and group based program. Each session lasts 90 minutes. Sessions occur approximately every other week.
  Arms: Healthy Thinking in Teens
Other: Advanced Diabetes Education. — 9 sessions. Manualized and group based program. Each session lasts 90 minutes. Sessions occur approximately every other week.
  Arms: Advanced Diabetes Education

SUMMARY:
Adolescents with type 1 diabetes are at increased risk for depressive symptoms, poor coping and problem-solving skills, poor regimen adherence, and negative diabetes-specific health outcomes. Although a handful of psychological interventions targeting adolescents' poor behavioral and emotional functioning demonstrate beneficial effects on disease management and outcomes, no prevention programs exist that equip adolescents with behavioral skills and cognitive strategies necessary to reduce these risks. Therefore, the proposed research will test whether a diabetes-specific adaptation of a resilience promoting, depression-prevention intervention for adolescents with type 1 diabetes will reduce both the risk of poor psychological functioning and the risk of negative health outcomes over time.

DETAILED DESCRIPTION:
1. Scope of Problem: Adolescents with type 1 diabetes (T1D) must balance a complex daily treatment regimen while also facing the emotional, social and academic demands of this developmental period. Not surprisingly, adolescents are at increased risk for anxiety and depressive symptoms, poor coping and problem-solving skills, poor regimen adherence, and negative diabetes-specific health outcomes. The mental and physical health risks of T1D add to its already staggering economic burden; the annual cost of diabetes in the United States for direct medical care exceeds $116 billion and individuals with diabetes have twice the healthcare costs of their peers without diabetes.

   A handful of psychological interventions targeting adolescents' poor behavioral and emotional functioning demonstrate beneficial effects on disease management and outcomes. However, no prevention programs exist that equip adolescents with behavioral skills and cognitive strategies shown to reduce both the risk of poor psychological functioning and the risk of negative health outcomes over time. Although none of the effective prevention programs developed for healthy youth have been adapted for adolescents with T1D, the Penn Resilience Program (PRP) is a viable candidate because it is a well-established prevention program shown to promote resilience and prevent depression. The current study will test a diabetes-specific adaptation of PRP for adolescents with T1D and fill a significant gap in the scientific literature.

   This study's significance lies not only in its focus on preventing depression, a prevalent, critical factor influencing diabetes-specific health outcomes, but also in its emphasis on ultimately preventing suboptimal glycemic control, a common, expensive, and dangerous problem in pediatric diabetes. Individuals with both depression and diabetes incur 4.5 times the health care costs as those with diabetes alone. The focus of the intervention on resilience promotion is innovative because of its potential to fundamentally change risk for depression and set adolescents on a trajectory toward improved adherence and health outcomes. Moreover, documenting the mechanisms of change that impact critical psychosocial and health outcomes in youth with T1D via a longitudinal, randomized, controlled design facilitates generalizability to other chronically ill populations given similar management demands on the individual and family, and associations with depression.
2. Summary of Procedures: Investigators will employ a randomized, controlled design and compare PRP T1D to a diabetes education intervention, (EI; developed by two CDE's, specifically focused on adolescent learning and adolescent needs) on resilience characteristics, depressive symptoms, adherence behaviors, and glycemic outcomes. Investigators will recruit 280 adolescents with T1D across two cities (Chicago and Cincinnati), measuring outcomes at baseline, post-intervention, and at five surveillance visits spanning an additional 24 months. All adolescents will participate in 9 sessions, lasting approximately 90 minutes each session. Assessments occur at baseline (0 months), post-intervention (4.5 months), and during the surveillance period (8, 12, 16, and 28 months).

   PRP T1D will be led by master's level graduate students enrolled in clinical psychology PhD programs. EI will be led by CDE nurses. This EI group is preferable to either untreated control or wait-list control groups as it allows for the experimental control of attention, peer group sessions, and dose on treatment outcomes. Both program leaders will receive over 20 hours of training in the program they are leading.

   Data Collection and Measures. Measures assess two primary outcomes (depressive symptoms and glycemic control) and two mechanisms of change (resilience and adherence). Assessments occur at baseline, post-intervention (4.5 months), and 4 surveillance visits (8, 12, 16, and 28 months). To keep participant burden at a manageable level and to increase retention rate, all eligible families will be invited to complete the questionnaires on a secured web-site that they can access while with the research study staff, or while at home, work, in a public library or while in clinic. Investigators will use the SNAP Survey Software system, which allows for electronic completion of surveys with data directly transferred to data management software in a HIPAA-protected framework. The SNAP software eliminates the need for manual data entry, reducing the risk of missing data as well as reducing the risk of violating the confidentiality of the data.

   Hemoglobin A1c will be collected via a small sample of blood and sent to a central laboratory. The Diabetes Diagnostic Laboratory at the University of Missouri (http://www.diabetes.missouri.edu/)will be used. This laboratory served as the reference laboratory for the DCCT and NHANES III and IV studies. They have extensive experience serving as a central laboratory for A1c values.

   Continuous glucose monitoring (CGM; iPro sensor and transmitter by Medtronic) will assess glycemic variability. The certified diabetes educator (CDE) or study physician will assist each participant with the insertion and calibration of the device. For this study, adolescents will be blinded to the CGM values for safety reasons; we do not want participants adjusting insulin levels or dietary intake based on sensor readings. Adolescents will wear the sensor and transmitter for 3 days. After use, the sensor/transmitter will be collected by the research team via a pre-paid mailing container. Once the transmitter is returned, the data are downloaded to study computers, typically with 290 values per day. Investigators then calculate three indicators of glycemic variability: SD of the mean of the sensor values, mean amplitude of glycemic excursions (MAGE), and percentage of time spent within glucose ranges. The amount of time spent "within target" (values between 70 and 180), "below target" (values below 70), and "above target" (values above 180) will be calculated. All three indicators are well-established metrics of glycemic variability.

   Enhancing Treatment Fidelity. Per the NIH Behavior Change Consortium,27 a randomized, controlled design is the most effective mechanism for finding treatment effects. Further, it is vital to insure all interventions are delivered as proposed and participants receive the same treatment dose within and across the intervention conditions. To achieve this, Investigators will make uniform reminder calls, use treatment manuals, and interventionists will meet every other week with the study PIs for group supervision to discuss relevant topics, problem areas, and plans for future sessions. Sessions will be audio taped so relevant points can be discussed in supervision. Ratings of audiotapes will be conducted by the PIs for 25% of the sessions, based on a list of key components.

   Frequent staff trainings is the key to delivering interventions as intended and to prevent drift. Therefore, staff training will occur twice annually in years 1-3 and once annually in years 4-5. Study PIs will coordinate the trainings which will be delivered collectively by the PIs and co-investigators. Training will cover delivery of the prevention program, coordinator activities (e.g., processing of blood samples for A1c), and treatment fidelity.
3. Risks: The risks in this study should be minor as many of the intervention components have been employed previously in research and clinical settings with minimal adverse events. The risks that come along with any study in which emotional and behavioral factors are discussed include the possibility of discomfort when completing questionnaires and during discussions in the intervention sessions. Further, given the nature of diabetes management, stress or patient-parent conflict may occur when uncontrolled blood sugars are documented. The research staff is trained to identify such distress or discomfort early and provide support in the intervention. Patients agreeing to participate in the studies will experience the usual risks associated with the treatment of type 1 diabetes: the most significant risk is hypoglycemia, which is present for all patients undergoing treatment for diabetes with insulin.

Another risk associated with this study is the threat to privacy and confidentiality if the secured website is somehow breached. However the SNAP software system and the secured web-site has been reviewed and approved by CMH's IT officers (Ron Isbell and Jason Ruprecht) and CMH's PHI officer (Valerie Witmer), and the PI has been using this secured website in another study without difficulties. Participants will access the questionnaires through the secured web-site and each participant will be assigned a unique study ID code number. Names, initials or other identifying information will not be used on any of the measures.

There may be other unknown risks for which investigators will monitor. An additional risk is the potential threat to privacy and confidentiality. Investigators believe that these represent minimal risks as defined by the DHHS office of Human Research Protection.

ELIGIBILITY:
Inclusion Criteria:

Study participants will meet the following inclusion criteria:

* 14-18 years old,
* diagnosis of T1D according to ADA criteria for at least 1 year,
* daily insulin dosing of at least 0.5 units per kilogram per day,
* fluent in English, and
* provide assent to participate.

Exclusion Criteria:

* other chronic, physical disease or condition except for celiac or thyroid disease,
* diagnosis of major depressive disorder determined at screening visit,
* current treatment with an antidepressant,
* diagnosis of major mental disorder (e.g., bipolar disorder, thought disorder, anorexia nervosa),
* diagnosis of developmental disorder (e.g., mental retardation, autism, asperger's), or ward of the state.

Adolescents must have established T1D, uncomplicated by other chronic diseases so any observed changes in glycemic control during the study cannot be attributed to other diseases or to endogenous insulin production seen in the 'honeymoon' period.28 Adolescents cannot have a diagnosis of major depressive disorder because that diagnosis warrants more intensive intervention. Further, adolescents cannot be on antidepressant medication treatment at the time they start the trial because it may impact psychological outcomes and cause unmeasured treatment effects. Finally, adolescents need to be without developmental or learning problems as that may make participation difficult, especially in a group format.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-09 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Depressive symptoms from baseline to post intervention and change in Depressive symptoms over the two year study period. | baseline, 4.5 months, 8.5 months, 12.5 months, 16.5 months, and 28.5 months
  Investigators expect that Depressive symptoms will change over time. Specifically, it is expected that depressive symptoms will not increase and may even decrease in the Healthy Thinking in Teens arm, whereas depressive symptoms will increase in the Advanced Diabetes Education arm.

SECONDARY OUTCOMES:
Change in Glycemic Control from baseline to post-intervention and change in Glycemic Control over time during the two year study period. | baseline, 4.5 months, 8.5 months, 12.5 months, 16.5 months and 28.5 months
  Hemoglobin A1C. Investigators expect that Hemoglobin A1C will change over time. Specifically, it is expected that Hemoglobin A1c will increase more in the Advanced Diabetes Education Arm than it will in the Healthy Thinking in Teens arm.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Weissberg-Benchell, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Shapiro JB, Bryant FB, Holmbeck GN, Hood KK, Weissberg-Benchell J. Do baseline resilience profiles moderate the effects of a resilience-enhancing intervention for adolescents with type I diabetes? Health Psychol. 2021 May;40(5):337-346. doi: 10.1037/hea0001076. PMID 34152787
- [Derived] Hood KK, Iturralde E, Rausch J, Weissberg-Benchell J. Preventing Diabetes Distress in Adolescents With Type 1 Diabetes: Results 1 Year After Participation in the STePS Program. Diabetes Care. 2018 Aug;41(8):1623-1630. doi: 10.2337/dc17-2556. Epub 2018 Jun 19. PMID 29921624